CLINICAL TRIAL: NCT00076869
Title: A Multicenter, Open, Noncomparative Study to Estimate the Safety, Tolerability, and Efficacy of MK0991 in Combination With Amphotericin B, Lipid Formulations of Amphotericin B, or Azoles in the Treatment of Invasive Aspergillus Infection in Adults Who Are Refractory to or Intolerant of Standard Therapy
Brief Title: MK0991 in Combination With Standard Antifungal Agent(s) for the Treatment of Salvage Invasive Aspergillosis (0991-037)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0991-037; Formally-0121FI; 2006_400
Record Dates: First submitted 2004-02-05; First posted 2004-02-06 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Aspergillosis
Keywords: Definite or probable Invasive Aspergillosis either refractory or intolerant to prior antifungal treatment.
MeSH Terms: conditions — Aspergillosis | interventions — Caspofungin

INTERVENTIONS:
Drug: MK0991, caspofungin acetate
Drug: Comparator: amphotericin B
Drug: Comparator: lipid formulation of amphotericin B and/or azole

SUMMARY:
Invasive aspergillosis is a type of fungal infection typically identified in very sick patients (for example, patients with cancer or who have had a bone marrow or organ transplant). This study will seek to enroll patients (16 years of age or older) with invasive aspergillosis infections (involving organs or deep tissues) who are failing or could not tolerate standard antifungal therapy. Your doctor will make this determination based upon specific study criteria. Patients that fulfill all study criteria will be treated daily with both the investigational drug and another antifungal agent. The choice of the other agent is up to your doctor. This investigational drug is approved for the treatment of invasive aspergillosis by itself. The safety and efficacy of this investigational drug, in combination with other agents is not known.

DETAILED DESCRIPTION:
The duration of treatment is 12 months.

ELIGIBILITY:
* Patients must meet a specific definition of probable or definite invasive aspergillosis and be considered to have failed or be intolerant of standard antifungal therapy.
* The patient must be at least 16 years old and if a woman of childbearing potential, must have a negative serum or urine pregnancy test sensitive to 25 IU hCG prior to enrollment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-01; Primary Completion 2004-09 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Tolerability.

SECONDARY OUTCOMES:
Clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Maertens J, Glasmacher A, Herbrecht R, Thiebaut A, Cordonnier C, Segal BH, Killar J, Taylor A, Kartsonis N, Patterson TF, Aoun M, Caillot D, Sable C; Caspofungin Combination Therapy Study Group. Multicenter, noncomparative study of caspofungin in combination with other antifungals as salvage therapy in adults with invasive aspergillosis. Cancer. 2006 Dec 15;107(12):2888-97. doi: 10.1002/cncr.22348. PMID 17103444